CLINICAL TRIAL: NCT05696249
Title: The Use of Pressure Sensors in Functional Assessment and Treatment of Low Back Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EK - 1499/22
Record Dates: First submitted 2023-01-08; First posted 2023-01-25 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Chronic Low-back Pain
Keywords: Intra-abdominal pressure; Biofeedback; Dynamometry

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with an OhmTrak device (Experimental): The intervention group will be equipped with an OhmTrak device for home self-therapy and instructed in its correct use at least 5 times a week.
  Interventions: Device: OhmTrak device.; Other: Outpatient Physiotherapy
- Group without an OhmTrak device (Other): The control group will receive identical outpatient therapy and instruction in self-therapy, except they will not have access to the OhmTrak device.
  Interventions: Other: Outpatient Physiotherapy

INTERVENTIONS:
Device: OhmTrak device. — All probands will undergo six-week outpatient therapy once a week. The intervention group will be equipped with an OhmTrak device for home self-therapy and instructed in its correct use at least 5 times a week.
  Arms: Group with an OhmTrak device
Other: Outpatient Physiotherapy — All probands will undergo six-week outpatient therapy once a week for an hour

SUMMARY:
The dissertation will focus on the possibilities of using pressure sensors during physiotherapy care. A single-blind randomized study will be conducted on a sample of at least 40 probands of working age with chronic LBP in the age range of 30-65 years. The following exclusive criteria are established: signs of serious spinal pathology (red flags), severe musculoskeletal trauma in the last year, vestibular, visual or neurological dysfunction affecting stability, ongoing pregnancy or breastfeeding, acute respiratory disease, cognitive dysfunction leading to misunderstanding of instructions and severe cardiac or internal disease. Inclusive and exclusive criteria will be evaluated by a rehabilitation doctor during a comprehensive examination before the start of therapy. All probands will undergo six-week outpatient therapy once a week. The intervention group will be equipped with an OhmTrak device for home self-therapy and instructed in its correct use at least 5 times a week. The control group will receive identical outpatient therapy and instruction in self-therapy, except they will not have access to the OhmTrak device. Before the start and at the end of the six-week therapy, all probands will be blindly evaluated for the quality of activation and use of intra-abdominal pressure with the DNS Brace device. At the same time, the Oswestry Disability Index questionnaire will be used to subjectively evaluate the probands before and after a series of therapies. The aim of the study is to demonstrate the possibility of using pressure sensors to improve the effect of physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patient with chronic Low Back Pain
* age range of 30-65 years.

Exclusion Criteria:

* signs of serious spinal pathology (red flags)
* severe musculoskeletal trauma in the last year
* vestibular, visual or neurological dysfunction affecting stability
* ongoing pregnancy or breastfeeding
* acute respiratory disease
* cognitive dysfunction leading to misunderstanding of instructions
* severe cardiac or internal disease

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Intra-abdominal pressure | six weeks
  Before the start and at the end of the six-weeks therapy, all probands will be blindly evaluated for the quality of activation and use of intra-abdominal pressure with the DNS Brace device.
Oswestry Disability Index, Version 2.1a | six weeks
  Before the start and at the end of the six-weeks therapy, all probands will fill in the Oswestry Disability Index questionnaire to evaluate their subjective state before and after a series of therapies. A score of zero equals no disability and a score of 100 is the maximum possible disability.

CONTACTS AND LOCATIONS:
Overall Officials: Alena Kobesova, prof., Study Director — Department of Rehabilitation and Sports Medicine, 2nd Faculty of Medicine and FN Motol
Locations (1):
- Centrum Pohybove Medicina Pavla Kolare a.s., Prague, Czechia

IPD SHARING:
Plan to Share IPD: No